CLINICAL TRIAL: NCT03985462
Title: Autologous Very Small Embryonic-like Stem Cells(VSELs) for Premature Ovarian Failure
Brief Title: Very Small Embryonic-like Stem Cells for Ovary
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Policy changes have contributed to the failure to carry out smoothly
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Guangzhou Four-Leaf Clover HealthTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSEL-ovary
Record Dates: First submitted 2019-06-01; First posted 2019-06-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05

CONDITIONS: Stem Cell Transplant Complications; Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients with confirmed premature ovarian failure were divided into three groups, each group was injected with different numbers of VSEL cells, and the control group was injected with platelet-rich serum which is the cell solvent
Who Masked: Investigator
Masking Description: The number of patients enrolled and the number of injected cells were randomly selected by the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VSEL Max (Experimental): A total of 300,000 VSEL cells in 5 mL plate-rich plasma are injected into the bilateral fallopian tubes as a high dose group
  Interventions: Biological: very small embryonic-like stem cell
- VSEL Medium (Experimental): A total of 200,000 VSEL cells in 5 mL plate-rich plasma are injected into the bilateral fallopian tubes as a middle dose group
  Interventions: Biological: very small embryonic-like stem cell
- VSEL Mini (Experimental): A total of 100,000 VSEL cells in 5 mL plate-rich plasma are injected into the bilateral fallopian tubes as a low dose group
  Interventions: Biological: very small embryonic-like stem cell
- Control (No Intervention): 5 mL plate-rich plasma with no cells inside were injected into the bilateral fallopian tubes as a control group

INTERVENTIONS:
Biological: very small embryonic-like stem cell — Mononuclear cells were collected from peripheral blood of each patient using a machine, VSELs were isolated, and each group was injected according to different numbers after activation
  Other Names: VSEL
  Arms: VSEL Max; VSEL Medium; VSEL Mini

SUMMARY:
The aim of this study is the safety and efficacy of autologous very small embryonic-like stem cells(VSELs) to premature ovarian failure.

DETAILED DESCRIPTION:
Premature ovarian failure is diagnosed by blood femal hormones test of follicle stimulating hormone (FSH, > 40 IU/L)、luteinizing hormon (LH, > 40 IU/L)、estradiol (E2, > 100pg/mL) and/or amenorrhea before the age of 40. VSELs come from the patient's periperal blood, and will be injected in bilateral oviducts, followed-up by hormone testing and menstrual conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as premature ovarian failure by professional doctor.
* Those have clear abnormal sex hormone levels

Exclusion Criteria:

* Unmarried woman
* Suffering from other serious gynecological diseases or gynecological tumors
* Blood disease patients, thrombocytopenia or dysfunction, hypofibrinemia or anticoagulant therapy, long-term use of aspirin

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients are enrolled in this research
Enrollment: 0 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Concentration of Blood female hormones level | 1 month after injection
  Check whether blood FSH, LH and E2 levels return to normal

SECONDARY OUTCOMES:
Concentration of Blood female hormones level | 6 months after injection
  Check whether blood FSH, LH and E2 levels return to normal
Incidence of amenorrhea | 6 months after injection
  Inquire about menstrual condition and exam ovarian blood supply by gynecological color ultrasound
Concentration of Blood female hormones level | 12 months after injection
  Check whether blood FSH, LH and E2 levels return to normal
Incidence of amenorrhea | 12 months after injection
  Inquire about menstrual condition and exam ovarian blood supply by gynecological color ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No